CLINICAL TRIAL: NCT04658238
Title: Associations of the Ocular Microbiome and the Immune System in Dry Eye Disease
Brief Title: Ocular Microbiome and Immune System in Dry Eyes
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Stiftung OPOS (Unknown); Fondation Bertarelli (Unknown)
Responsible Party: Sponsor
Other Study IDs: BASEC 2020-00775
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Dry Eye Disease
Keywords: microbiome; immune system
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA isolated from swabs frozen conjunctival tissue frozen tear fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dry eye disease: Patients with dry eye disease
  Interventions: Other: Ocular microbiome; Other: Ocular immune system
- Healthy controls: Healthy controls without dry eye disease
  Interventions: Other: Ocular microbiome; Other: Ocular immune system

INTERVENTIONS:
Other: Ocular microbiome — Taxonomical and functional characterization of the ocular microbiome
Other: Ocular immune system — Functional characterization of the tear fluid proteome, histology of conjunctival tissue and molecular assays

SUMMARY:
The primary objectives of this study are the characterization of the ocular microbiome as well as of the local immune system in participants with and without dry eye disease. Secondary objectives are the identification of differences in the ocular microbiome as well as in the immune system between participants with and without dry eye disease to ultimately find associations between the ocular microbiome and the immune system in dry eye disease.

DETAILED DESCRIPTION:
Although dry eye disease is considered to be one of the most common ocular surface diseases worldwide, treatment options are only very limited and severe side effects are common. However, recent studies showed that the ocular microbiome may be crucial for maintaining ocular surface homeostasis. Disruption of this homeostasis, called dysbiosis, may lead to inflammation that is a key component in the pathogenesis of dry eye disease. It has been suggested that bacteria are invasive in ocular mucosal tissue, thereby effectively hidden from clearance by the local immune system and rendering the inflammation chronic. Therefore, the investigators hypothesize that the ocular microbiome may induce changes in the mucosal immune system of the eye, which in turn may accelerate the development of dry eyes. Since there is a crucial role of both, the ocular microbiome and the local mucosal immune system, on several diseases, the overall aim of this project is to assess the associations of the mucosal immune system and the ocular microbiome in dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign informed consent
* 18 years of age or older

Exclusion Criteria:

* Not willing or able to sign informed consent
* Younger than 18 years
* Recent (3 month) history of use of systemic and/or topical antibiotics
* Usage of medical eye drops (Lacrycon and other moisturizing eye drops are allowed)
* Recent (3 month) history of ocular surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive ongoing recruitment of subjects attending routine follow-ups through the involved investigators in daily clinical practice at Department of Ophthalmology, Inselspital, Bern
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Ocular microbiome and local immune system in controls | At baseline
  Qualitative and quantitative characterization of the ocular microbiome and the local immune system in participants with no signs of dry eye disease. The primary variable for the characterization of the ocular microbiome is the identification of microbial taxa and the functional analysis of the identified taxa using eye swabs and conjunctival tissue samples. The primary variable for the characterization of the immune system is the identification of components of the ocular mucosal immune system (i.e. immune cells, anti- and proinflammatory cytokines) using conjunctival tissue samples and tear fluid. Baseline factors such as age, sex, BMI, medication, risk factors for dry eyes such as smoking and contact lenses may have an influence on the ocular microbiome.
Ocular microbiome and local immune system in patients | At baseline
  Qualitative and quantitative characterization of the ocular microbiome and the local immune system in participants with clinical signs of dry eye disease. For primary variable for characterization see Outcome 1. The variables for grading of dry eyes are tear film osmolarity, split lamp examination, tear secretion and subjective measurement by the "Ocular Surface Disease Index©" (OSDI©)" questionnaire.

SECONDARY OUTCOMES:
Differences of the ocular microbiome and the local immune system between patients and controls | At baseline
  Identification of differences of the ocular microbiome and the local immune system between patients and controls. The variables used for the differentiation of these two cohorts in terms of the microbiome are the relative abundances of identified microbial taxa and of corresponding functional features (i.e. genes and pathways) of the taxa. The variables used for the differentiation of the cohorts in terms of the immune system are quantitative values of cytokines and immune cells.
Correlations between the ocular microbiome and the local immune system | At baseline
  Identification of correlations between the ocular microbiome and the local immune system. For variables used see Outcome 3.

OTHER OUTCOMES:
Stability of the ocular surface microbiome | 3-6 months after baseline
  Sequential sample collection of eye swabs

CONTACTS AND LOCATIONS:
Overall Officials: Martin Zinkernagel, Prof. Dr. Dr., Principal Investigator — Department of Ophthalmology, Inselspital
Locations (1):
- Department of Ophthalmology, Inselspital, Bern, Switzerland

REFERENCES:
- [Derived] Sporri L, Studer JM, Kreuzer M, Rotzetter J, Scharer D, Largiader CR, Jaggi D, Zinkernagel MS, Zysset-Burri DC. Linking the microbiome to the complement system in geographic atrophy. NPJ Genom Med. 2026 Feb 2. doi: 10.1038/s41525-026-00550-7. Online ahead of print. PMID 41629364